CLINICAL TRIAL: NCT03675191
Title: The Effects of Orlistat/Phentermine Versus Placebo/Phentermine Treatment on Weight Loss and Vascular Function of Overweight Patients With Back Pain
Brief Title: Orlistat/Phentermine Versus Placebo/Phentermine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-Won Lee, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-2018-0210
Record Dates: First submitted 2018-08-28; First posted 2018-09-18 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Orlistat; Capsules; Phentermine

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled clinical trials (12 weeks)
  * orlistat (120mg, three times a day, within 1hour after meal) + phentermin (37.5mg, once a day, within 1hour after meal)
  * placebo (120mg, three times a day, within 1hour after meal) + phentermin (37.5mg, once a day, within 1hour after meal) The patients were divided into two groups: orlistat (120mg, three times a day), phentermine (37.5 mg, once a day) combined Group (N = 57), placebo (placebo, three times a day) and phentermine (37.5 mg, once a day) Group (N=57)
Who Masked: Participant, Care Provider, Investigator
Masking Description: The placebo pill is given to participants who are randomly assigned to the control group.
  Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orlistat (Experimental): Orlistat 120Mg Cap (120mg, three times a day, within 1hour after meal) combined with phentermine pill (37.5mg, once a day, within 1hour after meal)
  Interventions: Drug: Orlistat 120Mg Cap; Drug: Phentermine Pill
- placebo (Placebo Comparator): placebo (120mg, three times a day, within 1hour after meal) combined with phentermine pill (37.5mg, once a day, within 1hour after meal)
  Interventions: Drug: Phentermine Pill

INTERVENTIONS:
Drug: Orlistat 120Mg Cap — Drug,Orlistat 120Mg Cap, three times a day, within 1hour after meal
  Other Names: Lipidown Cap
  Arms: orlistat
Drug: Phentermine Pill — Drug,Phentermine Pill 37.5mg, both in two arms, one time a day, within 1hour after meal
  Other Names: Phentermine Pill 37.5mg

SUMMARY:
The prevalence of obesity is increasing worldwide and obesity is an important risk factor for cardiovascular disease. In addition, back pain has been increasing steadily due to sitting life, lack of exercise, wrong posture, and obesity. Recent studies found that obesity and back pain are common diseases and are closely related to each other. People with back pain have lower physical activity, which in turn leads to an weight gain and a deterioration in physical performance. Among the drugs used for obesity, orlistat has been approved for long-term use, and phentermine, the most commonly used drug, has been approved for short-term use. However, phentermine can increase blood pressure and pulse rate. Meanwhile, several studies have shown that orlistat, a pancreatic lipase inhibitor, lowers blood pressure and pulse rate and diminish LDL-cholesterol. Lowering LDL-C could lead to improved vascular endothelial function.

The investigators aimed to investigate the effect of orlistat and phentermine combination therapy on weight loss and improvement of vascular function compared to phentermine monotherapy in obese patients (BMI 27 kg/m2) with metabolic risk and back pain.

DETAILED DESCRIPTION:
The investigators aimed to investigate the effect of orlistat and phentermine combination therapy on weight loss and improvement of vascular function compared to phentermine monotherapy in obese patients (BMI 27 kg/m2) with metabolic risk and back pain.

Randomized placebo-controlled clinical trials (12 weeks), Patients: Obese patients (BMI 27 kg/m2) with metabolic risk and back pain

The patients were divided into two groups: orlistat (120mg, three times a day), phentermine (37.5 mg, once a day) combined Group (N = 57), placebo (placebo, three times a day) and phentermine (37.5 mg, once a day) Group (N=57).

Randomly assigned to each group at 1: 1, and allocation codes are generated using SAS (Ver. 9.2). The investigators provide orlistat and phentermine or placebo and phentermine. The investigators check physical measurement, blood test, questionnaire, blood pressure and pulse, body composition, FMD, heart rate variability test, in the first visit. The investigators check for changes in body weight, compliance, and side effects after 4 weeks and 8 weeks, respectively. After 12 weeks, the investigators re-check physical measurement, blood test, questionnaire, blood pressure and pulse, body composition, FMD, heart rate variability test.

ELIGIBILITY:
Inclusion Criteria:

* After a screening test, the characteristics of the trial were explained and then the patient voluntarily agreed to participate in the study and signed a consent form with IRB approval.
* Adults over 20 years of age at the time of obtaining consent
* A back pain score of 3 and a metabolic risk of a BMI greater than 27 kg / m2.
* Metabolic risk includes the following, according to the American Endocrinology Society (AACE) guidelines. (Diabetic stage, metabolic syndrome, type 2 diabetes, dyslipidemia, hypertension, cardiovascular disease, nonalcoholic fatty liver, polycystic ovary syndrome, obstructive sleep apnea, osteoarthritis, gastroesophageal
* In the case of a pregnant woman, pregnancy test is negative
* Patients who can understand and speak Korean
* Patients whose physicians approved to participate in the study
* Patients who are able to complete the study without participating in other intervention studies (drug, diet, exercise intervention studies) during the study period.
* Patients who agreed to contraception during the study

Exclusion Criteria:

1. Persons who are contraindicated for Phentermine Sympathomized excitable amines sensitive patients or patients with specific qualities Progressive arteriosclerosis patients Patients with symptomatic cardiovascular disease When there is pulmonary hypertension or heart valve disease A patient with hyperthyroidism A patient with glaucoma Patients who are extremely anxious or excited mentally person who had history of drug abuse Patients taking other central nervous system stimulants or those 14 days after the administration of MAO inhibitors (MAOIs)
2. Persons who are contraindicated for Orlistat Patient with chronic malabsorption syndrome or patient who stops secretion of juice Patients with hypersensitivity to this or this component
3. Uncontrolled hypertenstion (SBP>180mmHg or DBP >120mmHg)
4. Under taking anti-diabetics or fasting blood glucose >=200mg/dl
5. If your weight has decreased by more than 5 kg in the last 3 months
6. (AST or ALT> 3 times the normal value) or kidney disease (serum creatinine> 2.0 mg / dL)
7. Patients taking other clinical trial drugs
8. Patients taking other appetite suppressants within the last 30 days
9. Acute infectious diseases such as pneumonia, acute enteritis, and acute urinary tract infections
10. If you are participating in other clinical trials
11. Those who are deemed unsuitable for participating in this study by the researcher

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Body mass index changes | 12weeks
  Body mass index in kg/m2.
Vascular function changes | 12weeks
  Vascular function will be assessed using the flow mediated dilatation (%).

SECONDARY OUTCOMES:
Back pain | 12weeks
  Assessments using a Visual Analog Score for pain Visual Analog Scale (total score 10, minimum;0, no pain, maximum; 10, severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwon YJ, Lee H, Nam CM, Chang HJ, Yoon YR, Lee HS, Lee JW. Effects of Orlistat/Phentermine versus Phentermine on Vascular Endothelial Cell Function in Obese and Overweight Adults: A Randomized, Double-Blinded, Placebo-Controlled Trial. Diabetes Metab Syndr Obes. 2021 Mar 2;14:941-950. doi: 10.2147/DMSO.S300342. eCollection 2021. PMID 33688228